CLINICAL TRIAL: NCT01384214
Title: Pilot Study of the Effect of Botulinum Toxin Type A Treatment on Swallowing in Patients With Cervical Dystonia
Brief Title: Effect of Botulinum Toxin Type A on Swallowing in Patients With Cervical Dystonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Vice President Medical Affairs, Allergan, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedAff-BTX-0716
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Torticollis
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): botulinum toxin Type A
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — 750 U at Visit 1
  Other Names: Dysport®

SUMMARY:
The purpose of this study is to evaluate swallowing efficiency in patients with cervical dystonia following treatment with botulinum toxin Type A.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervical dystonia
* Successfully completed Allergan study MedAff BTX-0616 with 16 weeks since last botulinum toxin Type A injection
* In need of additional botulinum toxin Type A injections

Exclusion Criteria:

* Surgery or spinal cord stimulation for cervical dystonia
* Previous injections of phenol or alcohol for cervical dystonia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Oropharyngeal Swallow Efficiency (OPSE) | Baseline, Week 2

SECONDARY OUTCOMES:
Toronto Western Spasmodic Torticollis Scale (TWSTRS) Total Score | Week 4
Physician Assessment of Cervical Dystonia Severity | Week 4
Global Assessment of Benefit by Physician | Week 4
Global Assessment of Benefit by Patient | Week 4
Patient Visual Analog Assessment of Pain | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Zagreb, Croatia